CLINICAL TRIAL: NCT07013006
Title: Retrospective Study to Assess the Evolution of MRI or CT Lesions in Treated CNS Nocardiosis
Acronym: CENOCIM
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP250649
Record Dates: First submitted 2025-05-30; First posted 2025-06-10 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Nocardiosis
Keywords: Nocardiosis; Nocardia spp.; Radiological monitoring; Cerebral involvement
MeSH Terms: conditions — Nocardia Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patient suffering from cerebral nocardiosis defined by the presence of compatible clinical and radiological signs associated with the detection of Nocardia spp. in a biological sample (cerebral or extra-cerebral) between 01/01/2004 and 01/12/2024 with data collection that may continue 12 months after the end of treatment.
  Interventions: Other: Collection of data from the patient's medical file

INTERVENTIONS:
Other: Collection of data from the patient's medical file — Collection of data from the patient's medical file.

SUMMARY:
Nocardiosis is a rare infection caused by bacteria of the genus Nocardia spp. It primarily affects immunocompromised individuals, such as solid organ or hematopoietic stem cell transplant recipients, as well as individuals with anti-GM-CSF antibodies. The infection typically begins by inhalation, affecting the lungs, with frequent hematogenous spread to the brain and soft tissues. Cerebral involvement is present in 20 to 40% of cases, although 40% of patients remain neurologically asymptomatic.

Treatment consists of prolonged antibiotic therapy and, sometimes, surgical drainage for large or refractory abscesses. Mortality associated with cerebral involvement varies between 20 and 40%. Although radiological improvements are observed under treatment, the link between image changes and clinical prognosis remains uncertain. Regular radiological monitoring is recommended during and after treatment, although the expected evolution has not been described in the literature.

DETAILED DESCRIPTION:
Nocardiosis is a rare infection caused by bacteria of the genus Nocardia spp. It primarily affects immunocompromised individuals, such as solid organ or hematopoietic stem cell transplant recipients, as well as individuals with anti-GM-CSF antibodies. The infection typically begins by inhalation, affecting the lungs, with frequent hematogenous spread to the brain and soft tissues. Cerebral involvement is present in 20 to 40% of cases, although 40% of patients remain neurologically asymptomatic. Brain imaging is essential for diagnosis, with MRI often being preferred due to its sensitivity. Images often show multiple abscesses, but without sufficient specificity to differentiate nocardiosis from other pathogens. New MRI techniques could improve lesion characterization.

Treatment consists of prolonged antibiotic therapy and, sometimes, surgical drainage for large or refractory abscesses. Mortality associated with cerebral involvement varies between 20 and 40%. Although radiological improvements are observed under treatment, the link between image changes and clinical prognosis remains uncertain. Regular radiological monitoring is recommended during and after treatment, although the expected evolution has not been described in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Minor or adult patient with cerebral nocardiosis, defined by the presence of compatible clinical and radiological signs associated with the detection of Nocardia spp. in a biological sample (cerebral or extracerebral).
* With available imaging tests:

  * All patients with 3 brain imaging tests at the 3 stages of treatment: within 2 weeks of diagnosis, upon transition to maintenance treatment (3-6 weeks after the start of treatment), and at the end of treatment (between 1 month before and 1 month after the end of antibiotic treatment). MRI scans are preferred; in the absence of MRI images, contrast-enhanced CT scans will be included.
  * OR: any patient who has undergone an MRI and a contrast-enhanced CT scan within two weeks of diagnosis, with the two tests performed within 72 hours of each other.
  * OR: any patient with a multimodal brain MRI at any time during infection, preferably within one month of diagnosis.

Exclusion Criteria:

* Refusal or impossibility of information.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with cerebral nocardiosis and cared at an Assistance Publique -Hôpitaux de Paris hospital between 01/01/2004 and 01/12/2024.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Percentage reduction in cerebral nocardiosis lesions | 12 months
  Percentage reduction in cerebral nocardiosis lesions in patients with a favorable evolution and those with an unfavorable evolution at 12 months from diagnosis.

SECONDARY OUTCOMES:
Percentage of CT brain scans suggestive of cerebral nocardiosis | 12 months
  Percentage of CT brain scans finding abnormalities suggestive of cerebral nocardiosis, considering MRI as the gold standard for diagnosing cerebral nocardiosis.
Description of the variation in radiological presentation of cerebral nocardiosis lesions | 12 months
  Description of the variation in radiological presentation (number of abscesses, abscesses size, contrast uptake, vasculitic lesions, associated ventriculitis) according to the patient's background (transplantation, anti-GM-CSF antibodies, allogeneic CSH graft, others).
Percentage of cerebral vasculitis lesions | 12 months
  Percentage of cerebral vasculitis lesions on brain MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Margaux MD Garzaro, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Olivier MD, PhD Lortholary, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (13):
- France (13):
  - Hôpital Avicenne, Bobigny
  - Hôpital Ambroise-Paré, Boulogne-Billancourt
  - Hôpital Beaujon, Clichy
  - Hôpital Mondor, Créteil
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Hôpital Saint-Louis- Hôpital Lariboisière, Paris
  - Hôpital Armand-Trousseau, Paris
  - Hôpital Saint-Antoine, Paris
  - Hôpital Pitié-Salpêtrière, Paris
  - Hôpital Cochin, Paris
  - Hôpital Européen Georges-Pompidou, HEGP, Paris
  - Hôpital Necker-Enfants Malades, Paris
  - Hôpital Bichat - Claude-Bernard, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Averbuch D, De Greef J, Dureault A, Wendel L, Tridello G, Lebeaux D, Mikulska M, Gil L, Knelange N, Zuckerman T, Roussel X, Robin C, Xhaard A, Aljurf M, Beguin Y, Le Bourgeois A, Botella-Garcia C, Khanna N, Van Praet J, Kroger N, Blijlevens N, Ducastelle Lepretre S, Ho A, Roos-Weil D, Yeshurun M, Lortholary O, Fontanet A, de la Camara R, Coussement J, Maertens J, Styczynski J; European Study Group for Nocardia in Hematopoietic Cell Transplantation. Nocardia Infections in Hematopoietic Cell Transplant Recipients: A Multicenter International Retrospective Study of the Infectious Diseases Working Party of the European Society for Blood and Marrow Transplantation. Clin Infect Dis. 2022 Aug 24;75(1):88-97. doi: 10.1093/cid/ciab866. PMID 34596213
- [Background] Lebeaux D, Freund R, van Delden C, Guillot H, Marbus SD, Matignon M, Van Wijngaerden E, Douvry B, De Greef J, Vuotto F, Tricot L, Fernandez-Ruiz M, Dantal J, Hirzel C, Jais JP, Rodriguez-Nava V, Jacobs F, Lortholary O, Coussement J; European Study Group for Nocardia in Solid Organ Transplantation; European Study Group for Nocardia in Solid Organ Transplantation. Outcome and Treatment of Nocardiosis After Solid Organ Transplantation: New Insights From a European Study. Clin Infect Dis. 2017 May 15;64(10):1396-1405. doi: 10.1093/cid/cix124. PMID 28329348